CLINICAL TRIAL: NCT00048152
Title: A Randomized, Open-label Study Comparing the Effects of Low-dose Cyclosporine vs Cyclosporine Withdrawal on Renal Function in Kidney Transplant Patients Treated With CellCept and Daclizumab
Brief Title: A Study to Assess Use of Zenapax (Daclizumab) and CellCept (Mycophenolate Mofetil) to Improve Kidney Function in Kidney Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M67005
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Adrenal Cortex Hormones; Cyclosporine; Daclizumab; Mycophenolic Acid

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Corticosteroids; Drug: Neoral; Drug: Zenapax; Drug: mycophenolate mofetil [CellCept]
- 2 (Experimental)
  Interventions: Drug: Corticosteroids; Drug: Neoral; Drug: Zenapax; Drug: mycophenolate mofetil [CellCept]
- 3 (Experimental)
  Interventions: Drug: Corticosteroids; Drug: Neoral; Drug: mycophenolate mofetil [CellCept]

INTERVENTIONS:
Drug: Corticosteroids — As prescribed
Drug: Neoral — Low dose (target trough level 50-100ng/mL)
  Arms: 1; 2
Drug: Neoral — Standard dose (target trough level 150-300ng/mL)
  Arms: 3
Drug: Zenapax — 2mg/kg iv first dose, then 1mg/kg every 2 weeks
  Arms: 1; 2
Drug: mycophenolate mofetil [CellCept] — 1g po bid

SUMMARY:
This study will compare kidney function in kidney transplant patients following treatment with various combinations of Zenapax, CellCept, corticosteroids, and Neoral (Cyclosporine). The anticipated time on study treatment is 6-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients greater than 18 years of age
* recipients of primary kidney transplant
* single-organ recipients (kidney only)

Exclusion Criteria:

* previous treatment with Zenapax
* history of malignancy (except localized skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2000-12; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Renal function (as measured by GFR) | 12 months post-transplant

SECONDARY OUTCOMES:
Patient and graft survival \n | 12 months post-transplant
Proportion of patients with biopsy-proven rejection; treatment failure. | 6 and 12 months post-transplant
AEs, OIs, malignancies, deaths | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (35):
- United States (8):
  - Birmingham, Alabama
  - San Francisco, California
  - Gainesville, Florida
  - Atlanta, Georgia
  - Livingston, New Jersey
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Falls Church, Virginia
- Australia (2):
  - Adelaide
  - Sydney
- Belgium (2):
  - Brussels
  - Leuven
- Canada (4):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Saskatoon, Saskatchewan
- Vandœuvre-lès-Nancy, France
- Germany (3):
  - Berlin
  - Hanover
  - Münster
- Mexico (2):
  - Mexico City
  - Monterrey
- Oslo, Norway
- Poland (2):
  - Warsaw
  - Wroclaw
- Spain (5):
  - Barcelona
  - Córdoba
  - Málaga
  - Santander
  - Valencia
- Sweden (2):
  - Gothenburg
  - Malmo
- United Kingdom (3):
  - Birmingham
  - Glasgow
  - Leicester